CLINICAL TRIAL: NCT01208766
Title: A Randomized Phase III Study to Compare Bortezomib, Melphalan, Prednisone (VMP) With High Dose Melphalan Followed by Bortezomib, Lenalidomide, Dexamethasone (VRD) Consolidation and Lenalidomide Maintenance in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Study to Compare VMP With HDM Followed by VRD Consolidation and Lenalidomide Maintenance in Patients With Newly Diagnosed Multiple Myeloma
Acronym: HO95
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Collaborators: European Myeloma Network B.V. (Network); Gruppo Italiano Malattie EMatologiche dell'Adulto (Other); DSMM (Deutsche Studiengruppe Multiples Myelom) (Unknown); NMSG (Nordic Myeloma Study Group) (Unknown); Central European Myeloma Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOVON 95 MM; 2009-017903-28 (EudraCT Number); EMN02 (Other: European Myeloma Network)
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2026-01-06 (Actual); Status verified 2025-10

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma (Kahler's disease)
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Melphalan; Prednisone; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- R1: 4 cycles Bortezomib, Melphalan, Prednisone (VMP) (Active Comparator): All patients randomized to VMP treatment, will be treated with Bortezomib, Melphalan, Prednisone(VMP, 4 cycles) and will start intensification with VMP between 4 and 6 weeks after stem cell collection.
  Interventions: Drug: Bortezomib, Melphalan, Prednisone (VMP)
- R1: 1 (2) cycle(s) HDM (Experimental): All patients randomized to intensification with High Dose Melphalan will start intensification with HDM (in hospitals with a policy of double intensification, patients will be randomized between VMP, 1 HDM and 2 HDM) between 4 and 6 weeks after stem cell collection.
  Interventions: Drug: 1 or 2 cycle(s) HDM (High Dose Melphalan)
- R2: none (No Intervention): No consolidation, patients will continue to Lenalidomide maintenance.
- R2: 2 cycles of VRD (Experimental): In patients randomized to consolidation treatment, 2 cycles of Bortezomib, Lenalidomide,Dexamethasone (VRD) will start at 8 weeks after the end of the last course of VMP or HDM.
  Interventions: Drug: 2 cycles of Bortezomib, Lenalidomide, Dexamethasone (VRD)

INTERVENTIONS:
Drug: Bortezomib, Melphalan, Prednisone (VMP) — * Bortezomib _ 1.3 mg/m2 _ i.v. rapid infusion _ days 1,4,8,11,22,25,29,32
  * Melphalan _ 9 mg/m² _ p.o. _ days 1-4
  * Prednisone _ 60 mg/m² _ p.o. _ days 1-4
  Arms: R1: 4 cycles Bortezomib, Melphalan, Prednisone (VMP)
Drug: 1 or 2 cycle(s) HDM (High Dose Melphalan) — - Melphalan _ 100 mg/m² _ i.v. rapid infusion _ -3, -2*
  *Patients with renal insufficiency 100 mg/m2 only at day -3
  If a patient is randomized to receive 2 x HDM a second course of High Dose Melphalan may be administered between 2 and 3 months after the first course when the patient achieved at least PR.
  Arms: R1: 1 (2) cycle(s) HDM
Drug: 2 cycles of Bortezomib, Lenalidomide, Dexamethasone (VRD) — * Bortezomib _ 1.3 mg/m2 _ i.v. rapid infusion _ days 1,4,8,11
  * Lenalidomide _ 25 mg _ p.o. _ days 1-21
  * Dexamethasone _ 20 mg _ p.o. _ days 1,2,4,5,8,9,11,12
  Arms: R2: 2 cycles of VRD

SUMMARY:
Study phase: phase III

Study objective:

* Comparison of Bortezomib, Melphalan, Prednisone (VMP) with High Dose Melphalan followed autologous stem cell transplantation (ASCT)
* Comparison of Bortezomib, Lenalidomide, Dexamethasone(VRD) as consolidation versus no consolidation
* Comparison of single versus tandem high dose Melphalan with ASCT

Patient population: Patients with symptomatic multiple myeloma,previously untreated, ISS stages 1-3, age 18-65 years inclusive

Study design: Prospective, multicenter, intergroup, randomized

Duration of treatment: Expected duration of induction, stem cell collection and intensification is 6 - 9 months. Consolidation with VRD will last 2 months Maintenance therapy with Lenalidomide will be given until relapse. All patients will be followed until 10 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of symptomatic multiple myeloma stage I to III according to the International Staging System ISS (see appendix A), i.e. at least one of the CRAB criteria should be present;
* Measurable disease as defined by the presence of M-protein in serum or urine (serum M-protein> 10 g/l or urine M-protein > 200 mg/24 hours), or abnormal free light chain ratio;
* Age 18-65 years inclusive;
* WHO performance status 0-3 (WHO=3 is allowed only when caused by MM and not by comorbid conditions);
* Negative pregnancy test at inclusion if applicable;
* Written informed consent.

Inclusion for randomisation 1:

* WHO performance 0-2;
* Bilirubin and transaminases < 2.5 times the upper limit of normal values;
* A suitable stem cell graft containing at least 4 x 106 CD34+ cells/kg (or according to national guidelines).

Inclusion for randomisation 2:

* Bilirubin and transaminases < 2.5 times the upper limit of normal values;
* ANC >= 0.5 x 109/l and platelets > 20 x 10^9/l;
* Patient is able to adhere to the requirements of the Lenalidomide Pregnancy Prevention Risk Management Plan.

Exclusion Criteria:

* Known intolerance of Boron;
* Systemic AL amyloidosis;
* Primary Plasmacell Leukemia;
* Non-secretory MM;
* Previous chemotherapy or radiotherapy except local radiotherapy in case of local myeloma progression or corticosteroids maximum 5 days for symptom control;
* Severe cardiac dysfunction (NYHA classification II-IV);
* Significant hepatic dysfunction, unless related to myeloma;
* Patients with GFR <15 ml/min,
* Patients known to be HIV-positive;
* Patients with active, uncontrolled infections;
* Patients with neuropathy, CTC grade 2 or higher;
* Patients with a history of active malignancy during the past 5 years with the exception of basal carcinoma of the skin or stage 0 cervical carcinoma;
* Patients who are not willing or capable to use adequate contraception during the therapy (all men, all pre-menopausal women);
* Lactating women.

Exclusion for randomisation 1:

* Severe pulmonary, neurologic, or psychiatric disease;
* CTCAE grade 3-4 polyneuropathy during Bortezomib treatment;
* Allogeneic Stem Cell Transplantation (Allo SCT) planned;
* Progressive disease.'

Exclusion for randomisation 2:

* Progressive disease;
* Neuropathy, except CTCAE grade 1;
* CTCAE grade 3-4 polyneuropathy during Bortezomib treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2025-01 (Actual)

PRIMARY OUTCOMES:
For all registered patients: progression free survival (PFS) as defined by time from registration to progression or death from any cause (whichever occurs first). | end of trial (last patient last visit)
  For all registered patients: progression free survival (PFS) as defined by time from registration to progression or death from any cause (whichever occurs first).
For all patients included in R1; PFS as defined by time from randomization R1 to progression or death from any cause whichever comes first | end of trial (last patient last visit)
  For all patients included in R1; PFS as defined by time from randomization R1 to progression or death from any cause whichever comes first
For all patients included in R2; PFS as defined by time from randomization R2 to progression or death from any cause whichever comes first | end of trial (last patient last visit)
  For all patients included in R2; PFS as defined by time from randomization R2 to progression or death from any cause whichever comes first

SECONDARY OUTCOMES:
Overall survival measured from the time of registration /randomization R1/ randomization R2. Patients still alive or lost to follow up are censored at the date they were last known to be alive. | end of trial (last patient last visit)
  Overall survival measured from the time of registration /randomization R1/ randomization R2.
  Patients still alive or lost to follow up are censored at the date they were last known to be alive.
Toxicity | End of trial (last patient last visit)
  Toxicity
Response (PR, VGPR, CR and stringent CR), and improvement of response during the various stages of the treatment. | end of trial (last patient last visit)
  Response (PR, VGPR, CR and stringent CR), and improvement of response during the various stages of the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Sonneveld, Prof., Principal Investigator — Stichting Hemato-Oncologie voor Volwassenen Nederland
Locations (208):
- Australia (7):
  - AU-Brisbane-PAH, Brisbane
  - AU-Canberra-CANBERRAHOSPITAL, Canberra
  - AU-Melbourne-ALFRED, Melbourne
  - AU-Sydney-CONCORD, Sydney
  - AU-Sydney-NEPEAN, Sydney
  - Prince of Wales Hospital, Sydney
  - St George Hospital, Sydney
- Austria (3):
  - Krankenhaus d.Elisabethinen, Linz
  - Landeskrankenhaus Salzburg, Salzburg
  - AT-Vienna-HANUSCH, Vienna
- Belgium (11):
  - BE-Antwerpen Edegem-UZA, Antwerp
  - BE-Antwerpen-ZNASTUIVENBERG, Antwerp
  - BE-Haine-Saint-Paul-JOLIMONT, Haine-Saint-Paul
  - CHU Tivoli, La Louvière
  - BE-Liege-CHRCITADELLE, Liège
  - BE-Mons-AMBROISE, Mons
  - CHR Saint Joseph, Mons
  - BE-Roeselare-AZDELTA, Roeselare
  - RHMS, Saint-Ghislain
  - CH Wapi, Tournai
  - AZ Turnhout, Turnhout
- Czechia (6):
  - CZ-Brno-UHBRNO, Brno
  - Kralove-University Hospital Hradec Kralove, Hradec
  - CZ-Olomouc-FNOL, Olomouc
  - CZ-Ostrava-Poruba-FNO, Ostrava
  - University Hospital Plzen, Pilsen
  - University Hospital Kralovske Vinohrady, Prague
- Denmark (6):
  - DK-Aalborg-AALBORGUH, Aalborg
  - DK-Aarhus N-AUH, Aarhus
  - DK-Copenhagen-RIGSHOSPITALET, Copenhagen
  - DK-Herlev-HERLEV, Herlev
  - DK-Odense-OUH, Odense
  - DK-Roskilde-ROSKILDE, Roskilde
- FI-Turku-TYKS, Turku, Finland
- GR-Athens-ALEXANDRA, Athens, Greece
- Hungary (2):
  - St. Istvan and St. Laszlo Korhaz Hospital, Budapest
  - Szeged University Hospital, Szeged
- Italy (64):
  - SS Antonio e Biogio, Alessandria
  - AOU Umberto I-Clinica di Ematologica, Ancona
  - Ospedale C. e G. Mazzoni-Ematologia, Ascoli Piceno
  - A.O.R.N. San G. Moscati, Avellino
  - Policlinico di Bari, Bari
  - Oaspedali Riuniti_Div di Ematologia, Bergamo
  - Instituto di Ematologia e Oncologia Medica, Bologna
  - Ospedale Generale Regionale_Div di Ema e Centro, Bolzano
  - Spedali Civili_U.O.Ematologia, Brescia
  - Pres Osp Di Summa, Brindisi
  - Presidio Osp R. Binaghi, Cagliari
  - Inst per la Ricerca e la Cura del Cancro Di, Candiolo
  - Ospedale Ferrarotto-Ema, Catania
  - Presidio ospedaliero dell'annunziata, Cosenza
  - OspedaleCivico S Croce e carle, Cuneo
  - Ospedali Riuniti di Foggia, Foggia
  - Azienda Ospedaliera San Antonio Abate, Gallarate
  - Azienda Ospedaliera Universitaria S. Martino_Clinica Ematologica, Genova
  - Azienda Ospedaliera Universitaria S. Martino_Ematologia 1, Genova
  - Azienda Ospedaliera Universitaria S. Martino_Ematologia 2, Genova
  - Università La Sapienza Polo Pontino, Latina
  - Ospedale A. Manzoni, Lecco
  - ASUR Regione Marche, Marche
  - IRST, Meldola
  - Azienda Ospedaliera Papardo, Messina
  - Policlinico Gaetano Martino, Messina
  - Osp Dell Angelo, Mestre
  - Istituto Nazionale dei Tumori-Ema, Milan
  - Ospedale Niguarda Cà Grande, Milan
  - Policlinico- servizio di Ematologia, Modena
  - Ospedale Cardarelli-ematologia e Trapianto di Midollo Osseo, Napoli
  - Ospedale Cardarelli-Sezione di Ematologia TERE, Napoli
  - Universita Federico II-Ema, Napoli
  - Università Amedeo Avogrado-Ospedale Maggiore, Novara
  - Ospedale San Francesco, Nuoro
  - Osp San Luigi Gonzaga-Pat med, Orbassano
  - Ospedaliera di Pavona_Ematologia e, Padua
  - Giaccone di Palermo, Palermo
  - Fondazione Maugeri, Pavia
  - Policlinico San Matteo, Pavia
  - Azienda Ospedaliera S. Maria della Misericordia, Perugia
  - AO Ospedali Riunti Marche Nord, Pesaro
  - Presidio Osp dello Spirito Santo, Pescara
  - Osp S Maria delle Croci_Ema, Ravenna
  - A.O. Bianchi Melacrino Morelli_Ops Riunti, Reggio Calabria
  - Azienda Ospedaliera S. Maria Nuova, Reggio Emilia
  - Ospedale Infermi, Rimini
  - Ospedale Oncologica Regionale, Rionero in Vulture
  - Azienda Osp S. Andrea, Roma
  - Inst Regina elena-SC Ema IFO, Roma
  - Osp. san Camillo Forlanini, Roma
  - Ospedale S Eugenio_Ema, Roma
  - Ospedale San Giovanni Addolorata, Roma
  - UC Biomedico_Divisione di Ematologia, Roma
  - Universita La Sapienza_Ospedale Umberto I, Roma
  - Istituto Clinico Humanitas, Rozzano
  - AOU Senese Policlinico S. Maria alle Scotte, Siena
  - PO SS Ann e S.G. Moscati-Ema, Taranto
  - St. Maria_Oncoematologia, Terni
  - San Giovanni Battista Le Molinette-Ema 1, Torino
  - San Giovanni Battista Le Molinette-Ema 2, Torino
  - AO Cardinale G. Panico, Tricase
  - AOU Ospedali Riuniti, Trieste
  - AOU S.Maria della Misericordia, Udine
- LU-Luxembourg-CHL, Luxembourg, Luxembourg
- Netherlands (59):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Alkmaar-NWZ, Alkmaar
  - NL-Almere-FLEVOZIEKENHUIS, Almere Stad
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amstelveen-AMSTELLAND, Amstelveen
  - NL-Amsterdam-AMC, Amsterdam
  - NL-Amsterdam-AVL, Amsterdam
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Apeldoorn-GELREAPELDOORN, Apeldoorn
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Assen-WZA, Assen
  - NL-Beverwijk-RKZ, Beverwijk
  - NL-Breda-AMPHIA, Breda
  - NL-Capelle a/d IJssel-YSL, Capelle aan den IJssel
  - NL-Delft-RDGG, Delft
  - NL-Deventer-DZ, Deventer
  - NL-Dirksland-VANWEELBETHESDA, Dirksland
  - NL-Doetinchem-SLINGELAND, Doetinchem
  - NL-Dordrecht-ASZ, Dordrecht
  - Nij Smellinghe, Drachten
  - NL-Ede-ZGV, Ede
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Emmen-SCHEPER, Emmen
  - NL-Enschede-MST, Enschede
  - NL-Geldrop-STANNA, Geldrop
  - NL-Goes-ADRZ, Goes
  - NL-Gorinchem-BEATRIX, Gorinchem
  - NL-Gouda-GROENEHART, Gouda
  - NL-Groningen-UMCG, Groningen
  - NL-Heerlen-ATRIUMMC, Heerlen
  - NL-Helmond-ELKERLIEK, Helmond
  - NL-Hilversum-TERGOOI, Hilversum
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Hoorn-DIJKLANDERHOORN, Hoorn
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Nijmegen-RADBOUDUMC, Nijmegen
  - NL-Roermond-LZR, Roermond
  - NL-Roosendaal-BRAVIS, Roosendaal
  - NL-Rotterdam-EMCDANIEL, Rotterdam
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Rotterdam-IKAZIA, Rotterdam
  - NL-Rotterdam-MAASSTADZIEKENHUIS, Rotterdam
  - NL-Rotterdam-SFG, Rotterdam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Spijkenisse-SPIJKENISSEMC, Spijkenisse
  - NL-Terneuzen-ZORGSAAM, Terneuzen
  - NL-Den Haag-HAGA, The Hague
  - NL-Tilburg-ETZ, Tilburg
  - NL-Utrecht-DIAKONESSENUTRECHT, Utrecht
  - NL-Utrecht-UMCUTRECHT, Utrecht
  - NL-Venlo-VIECURI, Venlo
  - NL-Winterswijk-SKBWINTERSWIJK, Winterswijk
  - NL-Zwolle-ISALA, Zwolle
- Norway (12):
  - Helse Sunnmore, Ålesund
  - Haukeland University Hospital, Bergen
  - Forde Central Hosiptal, Førde
  - Harstad University Hospital, Harstad
  - Sørlandet Hospital, Kristiansand
  - Levanger Hospital, Levanger
  - NO-Lørenskog-AKERSHUS, Lørenskog
  - NO-Oslo-OSLOUH, Oslo
  - Baerum hospital, Sandvika
  - NO-Stavanger-HELSESTAVANGER, Stavanger
  - NO-Tromsø-NORTHNOORWEGEN, Tromsø
  - NO-Trondheim-STOLAV, Trondheim
- Francisco Gentil, Lisbon, Portugal
- Sweden (18):
  - SE-Boras-SASBORAS, Borås
  - Eskilstuna Malar Hospital, Eskilstuna
  - Falun Hospital, Falun
  - Sahlgrenska University Hospital, Gothenburg
  - Hallands Hospital Halmstad, Halmstad
  - Helsingborg General Hospital, Helsingborg
  - Ryhov Hospital, Jönköping
  - Lidkoping Hospital, Lidköping
  - SE-Linköping-REGIONOSTERGOTLAND, Linköping
  - SE-Luleå-SUNDERBY, Luleå
  - SE-Lund-SUH, Lund
  - Orebro University Hospital, Örebro
  - SE-Stockholm-KAROLINSKAHUDDINGE, Stockholm
  - Sundsvall Hospital, Sundsvall
  - Uddevall Hospital, Uddevalla
  - Umea University Hospital, Umeå
  - SE-Uppsala-UPPSALAUH, Uppsala
  - Centrallasareltet Vaxjo, Vaxjo
- Switzerland (10):
  - CH-Aarau-KSA, Aarau
  - CH-Basel-USB, Basel
  - CH-Bellinzona-IOSI, Bellinzona
  - CH-Bern-INSEL, Bern
  - KS Graubunden, Chur
  - CH-Geneve (14)-HCUGE, Geneva
  - Kantonsspital Baselland, Liestal
  - CH-Luzern-LUKS, Lucerne
  - CH-St. Gallen-KSSG, Sankt Gallen
  - CH-Zürich-USZ, Zurich
- Turkey (Türkiye) (6):
  - Baskent University Hospital, Adana
  - Gazi University Hospital, Ankara
  - University Hospital Ankara, Ankara
  - Istanbul University Hospital, Istanbul
  - Ege University Hospital, Izmir
  - Erciyes University Hospital, Kayseri

REFERENCES:
- [Derived] Mai EK, Hielscher T, Bertsch U, Salwender HJ, Zweegman S, Raab MS, Munder M, Pantani L, Mancuso K, Brossart P, Beksac M, Blau IW, Durig J, Besemer B, Fenk R, Reimer P, van der Holt B, Hanel M, von Metzler I, Graeven U, Muller-Tidow C, Boccadoro M, Scheid C, Dimopoulos MA, Hillengass J, Weisel KC, Cavo M, Sonneveld P, Goldschmidt H. Predictors of early morbidity and mortality in newly diagnosed multiple myeloma: data from five randomized, controlled, phase III trials in 3700 patients. Leukemia. 2024 Mar;38(3):640-647. doi: 10.1038/s41375-023-02105-6. Epub 2023 Dec 7. PMID 38062124
- [Derived] Schmitz A, Brondum RF, Johnsen HE, Mellqvist UH, Waage A, Gimsing P, Op Bruinink DH, van der Velden V, van der Holt B, Hansson M, Andersen NF, Frolund UC, Helleberg C, Schjesvold FH, Ahlberg L, Gulbrandsen N, Andreasson B, Lauri B, Haukas E, Bodker JS, Roug AS, Bogsted M, Severinsen MT, Gregersen H, Abildgaard N, Sonneveld P, Dybkaer K. Longitudinal minimal residual disease assessment in multiple myeloma patients in complete remission - results from the NMSG flow-MRD substudy within the EMN02/HO95 MM trial. BMC Cancer. 2022 Feb 5;22(1):147. doi: 10.1186/s12885-022-09184-1. PMID 35123422
- [Derived] Sonneveld P, Dimopoulos MA, Beksac M, van der Holt B, Aquino S, Ludwig H, Zweegman S, Zander T, Zamagni E, Wester R, Hajek R, Pantani L, Dozza L, Gay F, Cafro A, De Rosa L, Morelli A, Gregersen H, Gulbrandsen N, Cornelisse P, Troia R, Oliva S, van de Velden V, Wu K, Ypma PF, Bos G, Levin MD, Pour L, Driessen C, Broijl A, Croockewit A, Minnema MC, Waage A, Hveding C, van de Donk NWCJ, Offidani M, Palumbo GA, Spencer A, Boccadoro M, Cavo M. Consolidation and Maintenance in Newly Diagnosed Multiple Myeloma. J Clin Oncol. 2021 Nov 10;39(32):3613-3622. doi: 10.1200/JCO.21.01045. Epub 2021 Sep 14. PMID 34520219
- [Derived] Cavo M, Gay F, Beksac M, Pantani L, Petrucci MT, Dimopoulos MA, Dozza L, van der Holt B, Zweegman S, Oliva S, van der Velden VHJ, Zamagni E, Palumbo GA, Patriarca F, Montefusco V, Galli M, Maisnar V, Gamberi B, Hansson M, Belotti A, Pour L, Ypma P, Grasso M, Croockewit A, Ballanti S, Offidani M, Vincelli ID, Zambello R, Liberati AM, Andersen NF, Broijl A, Troia R, Pascarella A, Benevolo G, Levin MD, Bos G, Ludwig H, Aquino S, Morelli AM, Wu KL, Boersma R, Hajek R, Durian M, von dem Borne PA, Caravita di Toritto T, Zander T, Driessen C, Specchia G, Waage A, Gimsing P, Mellqvist UH, van Marwijk Kooy M, Minnema M, Mandigers C, Cafro AM, Palmas A, Carvalho S, Spencer A, Boccadoro M, Sonneveld P. Autologous haematopoietic stem-cell transplantation versus bortezomib-melphalan-prednisone, with or without bortezomib-lenalidomide-dexamethasone consolidation therapy, and lenalidomide maintenance for newly diagnosed multiple myeloma (EMN02/HO95): a multicentre, randomised, open-label, phase 3 study. Lancet Haematol. 2020 Jun;7(6):e456-e468. doi: 10.1016/S2352-3026(20)30099-5. Epub 2020 Apr 30. PMID 32359506
- [Derived] Gambella M, Omede P, Spada S, Muccio VE, Gilestro M, Saraci E, Grammatico S, Larocca A, Conticello C, Bernardini A, Gamberi B, Troia R, Liberati AM, Offidani M, Rocci A, Palumbo A, Cavo M, Sonneveld P, Boccadoro M, Oliva S. Minimal residual disease by flow cytometry and allelic-specific oligonucleotide real-time quantitative polymerase chain reaction in patients with myeloma receiving lenalidomide maintenance: A pooled analysis. Cancer. 2019 Mar 1;125(5):750-760. doi: 10.1002/cncr.31854. Epub 2018 Dec 18. PMID 30561775
- See also: Hovon website — http://www.hovon.nl